CLINICAL TRIAL: NCT04571060
Title: Double-Blind, Randomized, Placebo-controlled, Safety and Efficacy Trial of BHV-3500 (Zavegepant) Intranasal for the Acute Treatment of Migraine
Brief Title: Randomized Trial in Adult Participants With Acute Migraines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3500-301; C5301001 (Other: Pfizer)
Record Dates: First submitted 2020-09-11; First posted 2020-09-30 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Migraine
Keywords: Acute Migraine; Phonophobia; Photophobia; Nausea
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Participant.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zavegepant (Experimental): Participants administered a single intranasal dose of zavegepant 10 mg on occurrence of migraine with moderate or severe intensity within 45 days after randomization. The dose was administered using an Aptar Unidose System (UDS) liquid spray device.
  Interventions: Drug: Zavegepant
- Placebo (Placebo Comparator): Participants administered a single intranasal dose of zavegepant matching placebo on occurrence of migraine with moderate or severe intensity within 45 days after randomization. The dose was administered using an Aptar UDS liquid spray device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zavegepant — One dose of zavegepant
  Other Names: BHV3500
  Arms: Zavegepant
Drug: Placebo — One dose of matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of BHV-3500 (zavegepant) versus placebo in the acute treatment of moderate or severe migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has at least 1-year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, including the following:

   1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age
   2. Migraine attacks, on average, lasting about 4-72 hours if untreated
   3. Not more than 8 attacks of moderate to severe intensity per month within the last 3 months
   4. At least 2 consistent migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening period
   5. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening Period.
   6. Participants on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to screening visit and the dose is not expected to change during the course of the study.
   7. Participants with contraindications for use of triptans may be included provided they meet all other study entry criteria.
2. Male and Female participants ≥18 years of age.

Exclusion Criteria:

1. Participant with a history of HIV disease
2. Participant history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Participants with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
3. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however participants can be included who have stable hypertension and/or diabetes for at least 3 months prior to being enrolled).
4. Participants with major depressive episode within the last 12 months, major depressive disorder or any anxiety disorder requiring more than 1 medication for each disorder.
5. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or participants who have met DSM-V criteria for any significant substance use disorder within the past 12 months.
6. History of nasal surgery in the 6 months.
7. Evidence at screening of significant nasal conditions that may affect the administration or absorption of the nasal product (e.g. severe septum deviation, nasal deformity or blockage, inflammation, perforation, mucosal erosion or ulceration, polyposis, nasal trauma)
8. Participation in any other investigational clinical trial while participating in this clinical trial. Participation in a COVID-19 mRNA vaccine study (vaccine must be authorized under FDA emergency use authorization or approval) who are at least 30 days post last dose of the vaccine are permitted to be screened for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1978 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (93):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Coastal Clinical Research, LLC, An AMR Co., Mobile, Alabama
  - MD First Research, Chandler, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Axiom Research, LLC, Colton, California
  - Pharmacology Research Institute, Encino, California
  - eStudySite, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Clinical Research Institute, Los Angeles, California
  - Wr-Pri, Llc, Newport Beach, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - CT Clinical Research, Cromwell, Connecticut
  - Ki Health Partners, LLC dba New England Institute for Clinical Research, Stamford, Connecticut
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Meridien Research, Lake Mary, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - The Neurology Research Group, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Ideal Clinical Research, Pembroke Pines, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Clin-Med Research & Development, LLC, South Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - JSV Clinical Research Study, Inc., Tampa, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Northwest Clinical Trials Inc., Boise, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Collective Medical Research, Prairie Village, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Community Clinical Research Network, Marlborough, Massachusetts
  - Boston Neuro Research Center, South Dartmouth, Massachusetts
  - Medvadis Research Corporation, Waltham, Massachusetts
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Healthcare Research Network, Hazelwood, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Excel Clinical Research, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - Regional Clinical Research, Endwell, New York
  - Central New York Clinical Research, Manlius, New York
  - Fieve Clinical Research, Inc, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Montefiore Medical Center: Headache Center, The Bronx, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - PharmQuest LLC, Greensboro, North Carolina
  - PMG of Raleigh, LLC, Raleigh, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Hometown Urgent Care & Research/ Wellnow, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - OK Clinical Research LLC, Edmond, Oklahoma
  - Tekton Research, Inc., Yukon, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Union, Pennsylvania
  - MD First Research, Lancaster, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Donald J. Garcia, Jr, MD, PA, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Red Star Research LLC, Lake Jackson, Texas
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - Clinical Investigation Specialist, Inc., Kenosha, Wisconsin

REFERENCES:
- [Derived] Lipton RB, Croop R, Stock DA, Madonia J, Forshaw M, Lovegren M, Mosher L, Coric V, Goadsby PJ. Safety, tolerability, and efficacy of zavegepant 10 mg nasal spray for the acute treatment of migraine in the USA: a phase 3, double-blind, randomised, placebo-controlled multicentre trial. Lancet Neurol. 2023 Mar;22(3):209-217. doi: 10.1016/S1474-4422(22)00517-8. PMID 36804093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 90 sites in the United States.
Pre-assignment Details: A total of 1978 participants were enrolled, of which 1405 participants were randomized to zavegepant 10 mg dose group or placebo group. The randomization was stratified by the use of prophylactic migraine medication (yes or no). 573 participants were not randomized due to screen failure, lost to follow-up, non-compliance, or other reasons.
Groups:
- Zavegepant 10 mg: Participants administered a single intranasal dose of zavegepant 10 mg on occurrence of migraine with moderate or severe intensity within 45 days after randomization. The dose was administered using an Aptar Unidose System (UDS) liquid spray device.
Period: Overall Study
Arm/Group | Zavegepant 10 mg | Placebo
Started (Randomized) | 703 | 702
Treated | 629 | 653
Efficacy Analysis Set Participants (Treated participants who were randomized only once, had a migraine of moderate or severe pain intensity at the time of dosing, were treated with study drug, and had post-dose efficacy data) | 623 | 646
Completed | 622 (Participants who were randomized, received the study drug and completed the study.) | 653 (Participants who were randomized, received the study drug and completed the study.)
Not Completed | 81 | 49
Not completed — Lost to Follow-up from Randomization to Treatment | 17 | 9
Not completed — Never treated migraine | 47 | 36
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up from Treatment to End of Study | 7 | 0

BASELINE CHARACTERISTICS:
Population: Treated participants included enrolled participants who took the study drug (zavegepant or placebo).
Groups:
- Zavegepant 10 mg: Participants administered a single intranasal dose of zavegepant 10 mg on occurrence of migraine with moderate or severe intensity within 45 days after randomization. The dose was administered using an Aptar UDS liquid spray device.
- Total: Total of all reporting groups
Arm/Group | Zavegepant 10 mg | Placebo | Total
Number analyzed (Participants) | 629 | 653 | 1282
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (13.19) | 40.7 (13.46) | 40.8 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 551 | 1059
  Male | 121 | 102 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 114 | 146 | 260
  Not Hispanic or Latino | 515 | 507 | 1022
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 21 | 16 | 37
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 86 | 84 | 170
  White | 515 | 545 | 1060
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Prophylactic Migraine Medication Use at Randomization [Count of Participants; unit: Participants]
  Yes | 88 | 83 | 171
  No | 541 | 570 | 1111

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Pain at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the electronic clinical outcome assessment (eCOA) handheld device. Pain freedom was defined as pain level of none post-dose.
Time Frame: 2 hours post-dose
Population: Efficacy Analysis Participants included treated participants who were randomized only once, had moderate to severe pain at the time of dosing, and had non-missing, post-dose efficacy data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 23.6 [20.3 to 26.9] | 14.9 [12.1 to 17.6]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 8.8, 95% CI 2-sided [4.5 to 13.1]

2. Primary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia immediately before dosing using the eCOA handheld device. Symptom status (absent, present) was assessed post-dose using the eCOA handheld device separately for nausea, photophobia, and phonophobia. Freedom from MBS was defined as MBS reported at on-study migraine attack onset that was absent post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 39.6 [35.8 to 43.5] | 31.1 [27.5 to 34.7]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0012, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 8.7, 95% CI 2-sided [3.4 to 13.9]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Pain relief was defined as pain level of none or mild.
Time Frame: 2 hours post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 58.7 [54.9 to 62.6] | 49.7 [45.8 to 53.5]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0012, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 9.0, 95% CI 2-sided [3.6 to 14.5]

4. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 2 Hours Post-dose
Description: Functional disability level was assessed on a 4-point scale (normal function, mildly impaired, severely impaired, requires bedrest) using the eCOA handheld device. Normal function was defined as a functional disability level of normal post-dose in the subset of participants with functional disability (mildly impaired, severely impaired, requires bedrest) at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The Efficacy Analysis Participants with functional disability at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 570 | 593
Percentage of participants | 35.8 [31.9 to 39.7] | 25.6 [22.1 to 29.1]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 10.2, 95% CI 2-sided [5.0 to 15.5]

5. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 Hours to 24 Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 24 hours post-dose.
Time Frame: From 2 to 24 hours post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 40.6 [36.8 to 44.5] | 33.0 [29.3 to 36.6]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0048, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 7.6, 95% CI 2-sided [2.3 to 12.9]

6. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 Hours to 48 Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 48 hours post-dose.
Time Frame: From 2 to 48 hours post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 36.1 [32.3 to 39.9] | 29.6 [26.0 to 33.1]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0130, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 6.5, 95% CI 2-sided [1.4 to 11.7]

7. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 Hours to 24 Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain freedom was defined as pain level of none at 2 hours up to 24 hours post-dose.
Time Frame: From 2 to 24 hours post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 14.6 [11.8 to 17.4] | 9.8 [7.5 to 12.0]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0076, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 4.9, 95% CI 2-sided [1.3 to 8.5]

8. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 Hours to 48 Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain freedom was defined as pain level of none at 2 hours up to 48 hours post-dose.
Time Frame: From 2 to 48 hours post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 12.4 [9.8 to 14.9] | 8.7 [6.5 to 10.8]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0308, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 3.7, 95% CI 2-sided [0.3 to 7.1]

9. Secondary Outcome: Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose
Description: Phonophobia (sensitivity to sound) status was measured as absent or present in the eCOA handheld device. Freedom from phonophobia was defined as phonophobia absent post-dose in the subset of participants with phonophobia present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: Efficacy Analysis Participants with symptom of phonophobia present at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 407 | 425
Percentage of participants | 41.0 [36.3 to 45.8] | 32.7 [28.2 to 37.2]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0123, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 8.3, 95% CI 2-sided [1.8 to 14.9]

10. Secondary Outcome: Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose
Description: Photophobia (sensitivity to light) status was measured as absent or present in the eCOA handheld device. Freedom from photophobia was defined as photophobia absent post-dose in the subset of participants with photophobia present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: Efficacy Analysis Participants with symptom of photophobia present at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 558 | 585
Percentage of participants | 37.1 [33.1 to 41.1] | 28.5 [24.9 to 32.2]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0018, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 8.6, 95% CI 2-sided [3.2 to 14.1]

11. Secondary Outcome: Percentage of Participants With Pain Relief at 60 Minutes Post-dose
Description: as for outcome 3
Time Frame: 60 minutes post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 43.3 [39.4 to 47.2] | 37.3 [33.6 to 41.0]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0293, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 6.0, 95% CI 2-sided [0.6 to 11.4]

12. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 60 Minutes Post-dose
Description: Functional disability level was assessed on a 4-point scale (normal function, mildly impaired, severely impaired, requires bedrest) using the eCOA handheld device. Normal function was defined as a functional disability level of normal post-dose in the subset of participants with functional disability (mildly impaired, severely impaired, requires bedrest) present at on-study migraine attack onset.
Time Frame: 60 minutes post-dose
Population: The Efficacy Analysis Participants with normal function at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 570 | 593
Percentage of participants | 20.2 [16.9 to 23.5] | 15.5 [12.6 to 18.4]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0362, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 4.7, 95% CI 2-sided [0.3 to 9.1]

13. Secondary Outcome: Percentage of Participants With Pain Relief at 30 Minutes Post-dose
Description: as for outcome 3
Time Frame: 30 minutes post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 30.5 [26.9 to 34.1] | 20.3 [17.2 to 23.4]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 10.2, 95% CI 2-sided [5.5 to 15.0]

14. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 30 Minutes Post-dose
Description: as for outcome 4
Time Frame: 30 minutes post-dose
Population: The Efficacy Analysis Participants with normal function at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 570 | 593
Percentage of participants | 10.5 [8.0 to 13.0] | 6.1 [4.1 to 8.0]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p = 0.0059, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 4.4, 95% CI 2-sided [1.3 to 7.6]

15. Secondary Outcome: Percentage of Participants With Pain Relief at 15 Minutes Post-dose
Description: as for outcome 3
Time Frame: 15 minutes post-dose
Population: Efficacy analysis participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 623 | 646
Percentage of participants | 15.9 [13.0 to 18.8] | 8.0 [6.0 to 10.1]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at an alpha level of 0.05; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05; Stratified Percentage Difference = 7.8, 95% CI 2-sided [4.2 to 11.3]

16. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 15 Minutes Post-dose
Description: as for outcome 4
Time Frame: 15 minutes post-dose
Population: The Efficacy Analysis Participants with normal function at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 570 | 593
Percentage of participants | 3.3 [1.9 to 4.8] | 2.0 [0.9 to 3.2]

17. Secondary Outcome: Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose
Description: Participants who did not experience relief of their migraine headache at the end of 2 hours after dosing with study medication (and after the 2-hour assessments had been completed on the eCOA handheld device) were permitted to use the following rescue medications: aspirin, ibuprofen, acetaminophen up to 1000 mg/day (this includes Excedrin® Migraine), naproxen (or any other type of nonsteroidal anti-inflammatory drug), antiemetics (for example, metoclopramide or promethazine), or baclofen. The participant's use of rescue medication was recorded by the site on a case report form.
Time Frame: Through 24 hours post-dose
Population: Efficacy Analysis Participants were analyzed. Participants with rescue medication start date less than or equal to (≤) study drug start date + 1 day and missing rescue medication start time were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 620 | 643
Percentage of participants | 29.7 [26.1 to 33.3] | 35.8 [32.1 to 39.5]

18. Secondary Outcome: Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose
Description: Nausea status was measured as absent or present in the eCOA handheld device. Freedom from nausea was defined as nausea absent post-dose in the subset of participants with nausea present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The Efficacy Analysis Participants with symptom of nausea present at the time of dosing were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 380 | 405
Percentage of participants | 52.4 [47.3 to 57.4] | 50.9 [46.0 to 55.7]

19. Secondary Outcome: Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Pain relapse was defined as pain level of mild, moderate, or severe after 2 hours up to 48 hours post-dose in the subset of participants with pain level of none at 2 hours post-dose.
Time Frame: From 2 hours to 48 hours post-dose
Population: The Efficacy Analysis Participants with pain freedom at 2 hours post-dose were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 10 mg | Placebo
Number analyzed (Participants) | 147 | 96
Percentage of participants | 40.8 [32.9 to 48.8] | 35.4 [25.8 to 45.0]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from study drug dosing up to the end of the study (up to 55 days).
Description: Treated Participants included enrolled participants who took study therapy (zavegepant or placebo).
Groups:
- Placebo: Participants administered a single intranasal dose of zavegepant-matching placebo on occurrence of migraine with moderate or severe intensity within 45 days after randomization. The dose was administered using an Aptar UDS liquid spray device.
Arm/Group | Zavegepant 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/629 | 0/653
Serious Adverse Events (participants affected / at risk) | 0/629 | 0/653
Other Adverse Events (participants affected / at risk) | 129/629 | 31/653
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 10 mg (N=629) | Placebo (N=653)
Dysgeusia (Nervous system disorders) | 129 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT04571060/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04571060/SAP_001.pdf